CLINICAL TRIAL: NCT01419496
Title: Identifying Stat3-Dependent Chemotherapy Resistance Pathways in Relapsed AML
Brief Title: Study of Proteins in Promoting Chemotherapy Resistance in Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML12B1; COG-AAML12B1 (Other: Children's Oncology Group); AAML12B1 (Other: Children's Oncology Group); NCI-2011-02984 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with del(5q)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: protein expression analysis
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about cancer and development of drug resistance in patients.

PURPOSE: This research trial is studying proteins that may promote chemotherapy resistance in samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Investigate whether changes in prosurvival signaling occur by comparing activation of the signal transducer and activator of transcription-3 (Stat3) and Stat5 pathways in paired diagnostic and relapse samples.
* Investigate changes in leukemia cell responses to extrinsic cues from the environment change, using a bone marrow stromal-cell co-culture model of chemotherapy resistance.

OUTLINE: Cryopreserved samples are analyzed for Stat3 and Stat5 expression by flow cytometry and in vitro chemotherapy sensitivity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Paired diagnostic and relapsed cryopreserved samples from patients with acute myeloid leukemia

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in Stat3 and Stat5 in paired diagnostic and relapsed AML samples
Reduction in chemotherapy sensitivity by relapsed samples compared to diagnostic samples

CONTACTS AND LOCATIONS:
Overall Officials: Michele S. Redell, MD, PhD, Principal Investigator — Texas Children's Cancer Center